CLINICAL TRIAL: NCT04562688
Title: Care Improving Cognition for ADolescents on the Autism Spectrum (CICADAS)
Brief Title: Care Improving Cognition for ADolescents on the Autism Spectrum
Acronym: CICADAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PSC-0909-20
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Participants assigned to Arm A will engage in CICADAS app only for the first 16 weeks of the intervention period. After the completion of the first intervention period and the mid-intervention assessment (V3) visit, these participants will then be assigned to No-Contact (no active intervention) for the second 16 weeks of the intervention period.
  Interventions: Other: CICADAS only
- Arm B (Experimental): Participants assigned to Arm B will engage in PEERS + CICADAS for the first 16 weeks of the intervention period. After the completion of the first intervention period and the mid-intervention assessment (V3) visit, these participants will then be assigned to No-Contact (no active intervention) for the second 16 weeks of the intervention period.
  Interventions: Other: PEERS + CICADAS and then no-contact
- Arm C (Experimental): Participants assigned to Arm C will engage in PEERS + Active Comparator for the first 16 weeks of the intervention period. After the completion of the first intervention period and the mid-intervention assessment (V3) visit, these participants will then be assigned to No-Contact (no active intervention) for the second 16 weeks of the intervention period.
  Interventions: Other: PEERS + Active Comparator and then no-contact

INTERVENTIONS:
Other: CICADAS only — Participants completed baseline assessments and neuroplasticity-based targeted cognitive training (NB-TCT) exercises on a digital device for up to 40 hours through BrainHQ (Posit Science Corporation, San Francisco). The CICADAS app captures user-specific sensory and cognitive processing metrics through 10 brief computerized assessments; these data are used to guide and personalize the delivery of 13 NB-TCT exercises. The NB-TCT exercises are adaptive with the task difficulty adjusting on a trial-to-trial and session-by-session basis to the abilities of each individual. A second set of computerized assessments was administered following the intervention period. Participants had to log in to access these assessments and exercises using a study provided username that contained no personally identifiable information.
  Arms: Arm A
Other: PEERS + CICADAS and then no-contact — Participants will complete both PEERS and CICADAS study activities. Participants completed baseline assessments and neuroplasticity-based targeted cognitive training (NB-TCT) exercises on a digital device for up to 40 hours through BrainHQ (Posit Science Corporation, San Francisco). The CICADAS app captures user-specific sensory and cognitive processing metrics through 10 brief computerized assessments; these data are used to guide and personalize the delivery of 13 NB-TCT exercises. In addition, participants will be asked to attend weekly 1-hour group sessions led by a PEERS clinician. Each PEERS group session will consist of a minimum of 3 participants and will meet as a group using Zoom. PEERS teaches how to solve real-life social dilemmas, appraise affect and social contexts, and initiate and maintain conversations while receiving feedback from peers and clinicians. After 16 weeks, participant will crossover to No-Contact with no active intervention.
  Arms: Arm B
Other: PEERS + Active Comparator and then no-contact — Participants will complete both PEERS and Active Comparator study activities. Participants will engage in computerized, casual video games for a total of 40 hours. Participants will also complete the 10 sensory processing abnormalities (SPA) computerized assessments. In addition, participants will be asked to attend weekly 1-hour group sessions led by a PEERS clinician. Each PEERS group session will consist of a minimum of 3 participants and will meet as a group using Zoom. PEERS teaches how to solve real-life social dilemmas, appraise affect and social contexts, and initiate and maintain conversations while receiving feedback from peers and clinicians. After 16 weeks, participant will crossover to No-Contact with no active intervention.
  Arms: Arm C

SUMMARY:
This is a validation study to evaluate the acceptability, feasibility and impact of CICADAS (Care Improving Cognition for ADolescents on the Autism Spectrum), a clinician-assisted, digital application that aims to prime the brain to engage in flexible, adaptive long-term learning about social-emotional events through closed-loop technology.

DETAILED DESCRIPTION:
This study will employ an innovative and evidence-based digital intervention that includes ten digital assessments (CICADAS app) that will capture data on sensory processing abnormalities and associated cognitive deficits. We will leverage pilot data collected in adolescents with Autism Spectrum Disorder (ASD) and accumulate preliminary evidence for CICADAS app to function as 1) a stand-alone treatment; 2) a primer for PEERS (Program for the Education and Enrichment of Relationship Skills); 3) an enhancer for PEERS. This study will test CICADAS app in adolescents with ASD in a three-arm, active-controlled randomized crossover trial to document the acceptability and evaluate its potential as a stand-alone treatment, as a primer for PEERS, or as a treatment enhancer of PEERS.

ELIGIBILITY:
Inclusion Criteria:

1. Potential participant is between the age of 11 and 18 (inclusive) at the time of consent.
2. Potential participant has a clinical diagnosis of Autism Spectrum Disorder (ASD), as confirmed by medical/clinical records or standardized assessments/interviews (e.g., Autism Diagnostic Observation Schedule, 2nd Edition (ADOS-2) or Autism Diagnostic Interview - Revised (ADI-R)).
3. Potential participant has an IQ Score > 70 on the Wechsler Abbreviated Scale of Intelligence (WASI-II) or a comparable measure in medical/clinical records.
4. Potential participant has normal or corrected to normal vision (20/20 or better; self/parent-reported.
5. Potential participant has normal hearing (self/parent-reported).
6. Potential participant is a fluent English speaker, based on participant and/or parent/legal guardian self-report and as determined by the screening clinician, to ensure reasonable neuropsychological results on key assessments.
7. Potential participant has adequate sensorimotor capacity to perform the intervention and study activities, including visual capacity adequate to read from a computer screen or mobile device at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control and use a mobile device and/or computer, based on participant and/or parent/legal guardian self-report and as determined by the screening clinician and/or study team.
8. Potential participant must be clinically stable as a result of therapy or medication regimen for 4 weeks prior to enrolling into the study.
9. Potential participant has reliable access to the internet.

Exclusion Criteria:

1. Potential participant has history of psychotic disorders and/or seizure disorder and/or seizure episodes within the last 2 years.
2. Potential participant has a motor/perceptual handicap that prevents digital device use, as determined by the screening clinician and/or study team.
3. Potential participant has problems in performing assessments or comprehending or following spoken instructions, as determined by the screening clinician and/or study team.
4. Potential participant has medical illnesses/genetic syndromes deemed to interfere with participation in study activities and/or unstable and/or untreated conditions that may affect cognition, including substance abuse/dependence disorders, ongoing chemotherapy or other cancer treatment.
5. Potential participant has a history of head trauma, traumatic brain injury, or other neurological disorder that impairs cognition
6. Potential adult participant scores less than a 14 (75%) on the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC). Please note, this criteria applies only to adult participants, age 18, at the time of screening.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Digital Assessment Completion Rate | 16 weeks
  The completion rate for digital assessments will be evaluated.
NB-SCT Program Adherence | 16 weeks
  Program adherence based on percentage of sessions completed will be evaluated.
Post-Study Usability Ratings | 16 weeks
  The ratings on a post-study questionnaire that looks at program satisfaction, clarity, enjoyment, perceived benefits and ease of fit into schedule will be evaluated.
Reported Number of Adverse Effects | 16 weeks
  The reported number of adverse events due to program use will be evaluated.
Total number of participants who complete the intervention | 16 weeks
  The program completion rate will be evaluated.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) | 16 weeks and 32 weeks
  Assesses impairments in executive function across three composite indexes: Behavior Regulation, Emotional Recognition, and Cognitive Regulation.
Brain-Body Center Sensory Scales (BBCSS) | 16 weeks and 32 weeks
  Measures sensory vulnerabilities of auditory processing, visual processing, tactile processing, and eating and feeding behaviors.
Child Behavior Checklist (CBCL) | 16 weeks and 32 weeks
  Measure of behavioral and emotional functioning; subscales consistent with DSM-5 categories of Depressive, Anxiety, Somatic, Attention Deficit/Hyperactivity, Oppositional Defiant. and Conduct Problems.
Pediatric Qualify of Life Inventory (PedsQL) | 16 weeks and 32 weeks
  Measures health-related quality of life.
Repetitive Behavior Scale - Revised (RBS-R) | 16 weeks and 32 weeks
  Measures breadth of repetitive behavior with subscales: Stereotyped Behavior, Self-injurious Behavior, Compulsive Behavior, Routine Behavior, Sameness Behavior, and Restricted Behavior.
Social Responsiveness Scale, Second Edition (SRS-2) | 16 weeks and 32 weeks
  Measures severity of autism spectrum symptoms as they occur in natural social settings.
Social Skills Improvement System (SSIS) | 16 weeks and 32 weeks
  Assesses social skills, problem behaviors, and academic competence.
Flanker Task | 16 weeks and 32 weeks
  Test of selective attention and inhibitory control, in which participants are asked to indicate the target letter while ignoring an array of "flanking" congruent/incongruent letters.
SCAN-3:A Tests for Auditory Processing Disorders | 16 weeks and 32 weeks
  Screening for auditory processing difficulties Subtests: competing Words (dichotic listening tasks) and Filtered Words (speech processing when the signal is distorted or compromised by a poor acoustic environment).
Test of Adolescent Social Skills Knowledge (TASSK) | 16 weeks and 32 weeks
  Assesses treatment changes in adolescents' knowledge of social skills taught during PEERS.
Wisconsin Card Sorting Test (WCST) | 16 weeks and 32 weeks
  Neuropsychological test of set-shifting, the capability to show flexibility when exposed to changes in reinforcement.

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Lee, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States